CLINICAL TRIAL: NCT01315301
Title: Randomized Clinical Trial to Determine the Most Appropriate Time to Start HIV Treatment in HIV & TB Coinfected Adults Being Treated for Tuberculosis.
Brief Title: Optimal Time to Initiate Antiretroviral Therapy in HIV & TB Coinfected Adults Being Treated for Tuberculosis
Acronym: TB-HAART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Addis Ababa University (Other)
Responsible Party: Eleni Aklillu,PhD, Associate Professor, Karolinska Institutet, Stockholm, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SWE-2007-270
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Acquired Immunodeficiency Syndrome; Tuberculosis
Keywords: Efavirenz; Rifampicin; HAART; Anti Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm-A (Active Comparator): Immediate Treatment Group
  Interventions: Other: Comparison of different treatment strategies
- Arm-B (Active Comparator): Deferred Treatment Group-1
  Interventions: Other: Comparison of different treatment strategies
- Arm-C (Active Comparator): Deferred Treatment Group-2
  Interventions: Other: Comparison of different treatment strategies

INTERVENTIONS:
Other: Comparison of different treatment strategies — 600 mg efavirenz based HAART initiated one week after starting rifampicin based short course anti tuberculosis treatment.
  Other Names: Treatment
  Arms: Arm-A
Other: Comparison of different treatment strategies — 600 mg efavirenz based HAART initiated four weeks after starting rifampicin based short course anti tuberculosis treatment
  Other Names: Treatment
  Arms: Arm-B
Other: Comparison of different treatment strategies — 600 mg efavirenz based HAART initiated eight weeks after starting rifampicin based short course anti tuberculosis treatment.
  Other Names: Treatment
  Arms: Arm-C

SUMMARY:
Aim of the study is to determine optimal time to initiate anti-retroviral therapy in HIV/TB co-infected patients who recently started treatment for Tuberculosis by comparing immediate versus deferred initiation of HAART.

The study will address the following questions;

* Is it possible to reduce mortality rate and increase survival by early initiation of HAART during TB treatment with out compromising for adverse drug reaction, toxicity and immune reconstitution syndrome?
* What is the risk/ benefit ratio between immediate versus deferred initiation of HAART during TB treatment with respect to safety/efficacy of TB and HIV co-treatment?
* When is the most appropriate time to start HAART during TB treatment?

DETAILED DESCRIPTION:
The study intends to determine the optimal time to start ART by comparing three treatment strategies of ART initiation in HIV/TB co-infected patients. Four hundred fifty newly diagnosed HIV infected patients with active TB and CD4 cell count < 200 cells/mm3 will be prospectively recruited to be assigned randomly in parallel into one of the three treatment groups (n=150 in each group) and HAART will be started at different time points as described below with extensive counseling and adherence support.

* Arm-A (Immediate Treatment Group): Receipt of antiretroviral therapy one week after starting anti-TB treatment.
* Arm-B (Deferred Treatment Group-1): Antiretroviral therapy will be initiated at the 4th week of starting anti-TB treatment (in the middle of the intensive phase TB treatment).
* Arm-C (Deferred Treatment Group-2): Antiretroviral therapy will be initiated at the 8th week of starting anti-TB treatment (after completion of the intensive phase of TB treatment).

Study Design: Interventional, prospective, randomized, open-label three-armed trial with no placebo, Active control, parallel assignment, safety and efficacy study.

Study population: Previously untreated HIV-infected adult patients with TB and CD4 cell counts < 200/mm3 at the time of TB diagnosis.

Expected Total Enrollment = 450

Treatment: Patients will receive first-line preferred regimen for patients with TB and HIV coinfection (rifampicin containing short course TB treatment and efavirenz-containing HAART regimen. The intensive phase of anti-TB therapy consists of 2 months treatment with Rifampicin, Isoniazid, Pyrazinamide and Ethambutol followed by the continuation phase with Isoniazid and Rifampicin daily for 4 months under Directly Observed Therapy (DOTS). After the initiation of TB treatment, patients in Arm-A, Arm-B and Arm-C will start EFV-containing HAART regimen (efavirenz + Lamivudine (3TC) + Stavudine (d4T) after one week, in the middle(at 4th week) and at the end (8th week) of the intensive phase TB treatment respectively. Primar prophylaxis with cotrimoxazole will be offered to all patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ART naive HIV infected patients and age > 18 years old
* Newly diagnosed smear +ve PTB cases (abnormal CXR and at least one sputum sample +ve for AFB)
* Newly diagnosed smear -ve PTB cases (CXR consistent with active TB plus at least two sputum specimens negative for AFB and decision by the physician to treat for TB or smear negative for AFB but culture positive cases)
* Tissue biopsy or FNAC results consistent with the diagnosis of tuberculosis
* CD4 cell count < 200/mm3 at the time of TB diagnosis
* Residence in Addis Ababa, Ethiopia
* Ability to give signed written/thumb sign informed consent

Exclusion Criteria:

* Pregnancy and breast-feeding women
* Patients who received anti TB therapy with in the past two years
* Patients who have previous treatment experience with antiretroviral therapy
* Severely ill patients Karnofsky performance status score < 40
* Baseline Hgb < 8 gms/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
mortality | 24 weeks
  all cause mortality

SECONDARY OUTCOMES:
Tuberculosis-Immune Reconstitution Inflammatory Syndrome | 24 weeks
New AIDS defining clinical events | 24 weeks
Drug Induced Liver toxicity | 24 weeks
Virologic success | 24 weeks
  Proportion of patients with Virologic success defined as achieving a viral load of < 50 HIV-1 RNA copies/mL within 6 months of starting therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Aklillu, PhD, Study Director — Krolinska Institutet, Stockholm, Sweden; Wondwossen Amogne, MD, Principal Investigator — Addis Ababa University, Addis Ababa, Ethiopia
Locations (1):
- Tikur Anbessa (Black Lion) Hospital, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Amogne W, Aderaye G, Habtewold A, Yimer G, Makonnen E, Worku A, Sonnerborg A, Aklillu E, Lindquist L. Efficacy and Safety of Antiretroviral Therapy Initiated One Week after Tuberculosis Therapy in Patients with CD4 Counts < 200 Cells/muL: TB-HAART Study, a Randomized Clinical Trial. PLoS One. 2015 May 12;10(5):e0122587. doi: 10.1371/journal.pone.0122587. eCollection 2015. PMID 25966339